CLINICAL TRIAL: NCT04489823
Title: PARADIGM PARAvalvular Leak Closure With the Amplatzer Valvular Plug occluDer for Interventional Transcatheter Closure for PVL With Surgical bioloGical and Mechanical Heart Valve
Brief Title: PARADIGM: Amplatzer Valvular Plug for PVL Closure
Acronym: PARADIGM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10309
Record Dates: First submitted 2020-07-10; First posted 2020-07-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Paravalvular Aortic Regurgitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Paravalvular Leak Closure (Experimental): Includes all eligible subjects who undergo an AVP III implant attempt for treatment of significant paravalvular leakage with an echocardiographic severity grade of moderate or higher. This is a single arm study.
  Interventions: Device: AVP III

INTERVENTIONS:
Device: AVP III — Transcatheter closure of a paravalvular leak using AVP III

SUMMARY:
The Paradigm study is a prospective, multicenter, single arm study to demonstrate the safety and effectiveness of the Amplatzer Valvular Plug III (AVP III) as a treatment for clinically significant PVLs following surgical implant of a mechanical or biological heart valve implanted in the aortic or mitral position.

DETAILED DESCRIPTION:
PARADIGM is a prospective, international, multi-center, single arm study to demonstrate the safety and effectiveness of the AVP III for percutaneous, transcatheter closure of paravalvular leak (PVL) occurring after aortic or mitral valve replacement with a surgically-implanted mechanical or bioprosthetic valve. The study will be conducted at approximately 25 clinical sites in the US, Europe, and Canada. A total of 200 subjects with a clinically significant PVL will undergo an AVP III implant procedure for PVL closure. Pre-procedural Baseline and follow-up assessments at Discharge, 30 days, 6 months and 1 year will include echocardiography, physical examinations, lab measurements and questionnaires to assess PVL severity, prosthetic valve function, hemolytic anemia, heart failure symptoms, and quality of life. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is implanted with a mechanical or biological surgical valve in the aortic or mitral position
* Note: Subjects in European countries can only be implanted with a mechanical valve in the aortic or mitral position
* Subject has a clinically significant paravalvular leak with a severity grade of moderate or higher, associated with signs of heart failure and/or hemolysis necessitating recurring blood transfusions.
* Subject has one clinically significant PVL defect that can be closed with a single AVP III as assessed pre-procedurally
* Subject has provided written informed consent
* Subject is ≥18 years old

Exclusion Criteria:

* Subject has a rocking valve or extreme dehiscence of the prosthetic valve involving more than 40% of the sewing ring
* Subject's PVL(s) originates from a transcatheter aortic or mitral valve replacement, or from rapid deployment or sutureless surgical replacement valves
* Subject has a prosthetic aortic valve and prosthetic mitral valve which both have a clinically significant paravalvular leak.
* Subject who is hemodynamically unstable or who cannot undergo an elective procedure
* Subject with active endocarditis or other active infection
* Subject has within the last 6 months a previously documented intracardiac mass, vegetation, tumor, or thrombus which would interfere with placement of the AVP III
* Subject has inadequate vasculature for delivery of the AVP III
* Subject has unsuitable anatomy for PVL closure using the AVP III (such as a PVL associated with an abscess cavity or a pseudoaneurysmal sac) or anatomy where the AVP III would interfere with other intracardiac or intravascular structures (such coronary ostia)
* Subjects who are unable to receive intraprocedural anticoagulant therapy
* Pregnant or nursing subjects or subjects who plan pregnancy during the clinical investigation follow-up period.
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
* Life expectancy is less than 1 year in the opinion of the Investigator
* Incapacitated individuals, defined as persons with mental illnesses or handicaps that impair their ability to provide informed consent, or individuals without legal authority to provide informed consent.
* Individual who are currently participating in an investigational drug or device study that has not reached the primary endpoint or that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Paravalvular leak closure success rate (percent of subjects) | 30 Days
  * Successful transcatheter placement in the intended location without interference
  * Reduction in paravalvular regurgitation severity by ≥ two grades
  * Freedom from intra-procedural death
  * Freedom from unplanned transcatheter or surgical re-intervention through 30 days post-implant.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ruiz, M.D., Ph.D, Principal Investigator — Hackensack Meridian Health
Locations (24):
- United States (14):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Lenox Hill Hospital, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Canada (2):
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Institut de Cardiologie de Quebec (Hôpital Laval), Québec, Quebec
- Ospedale San Raffaele, Milan, Lombard, Italy
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands
- Gornoslaskie Centrum Medyczne im.prof. Leszka Gieca, Katowice, Silesian Voivodeship, Poland
- Spain (2):
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - Edinburgh Heart Centre, Edinburgh, Lothian
  - The Royal Sussex County Hospital, Brighton, Soeast
  - Papworth Hospital NHS Foundation Trust, Cambridge

IPD SHARING:
Plan to Share IPD: No